CLINICAL TRIAL: NCT00122395
Title: A Randomized Clinical Trial Regarding the Acceptability of an Audiotape Questionnaire for Intimate Partner Violence Screening in a Pediatric ED
Brief Title: Trial Regarding the Acceptability of Audiotape Intimate Partner Violence (IPV) Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004-5-3793
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2006-05-04 (Estimated); Status verified 2005-07

CONDITIONS: Domestic Violence
Keywords: Domestic violence; Screening; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Paper

INTERVENTIONS:
Behavioral: Screening via pen and paper
Behavioral: Screening via audiotape

SUMMARY:
The purpose of this study is to compare the safety, acceptability and ease of the administration of two screening methods, a pen and paper questionnaire and an audiotape with headsets, for screening for intimate partner violence in a pediatric emergency department (ED).

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a significant health problem, affecting 2 - 4 million women each year. Over half of the homes in which women are abused contain children, with 3.3 - 10 million children witnessing IPV each year. In 1998, the American Academy of Pediatrics (AAP) issued guidelines stating that "identifying and intervening on behalf of battered women may be one of the most effective means of preventing child abuse," and recommending that pediatricians perform routine IPV screening. Because of the substantial number of families seen in the emergency department (ED), this setting could provide an important site in which to implement universal screening. Exactly how to implement screening in this busy environment is unclear. One possible approach involves the use of an audiotape with a headset with a prerecorded screening questionnaire that prompts the respondent to circle "yes" or "no" answers on an otherwise blank sheet of paper. This method of screening has the potential benefits of:

* Providing a more private method of screening;
* Improving screening of women who cannot read well;
* Enhancing the rate of screening by removing the burden of screening from providers.

Comparison: Female caregivers in a pediatric ED will be randomized to answering domestic violence (DV) screening questions either via pen and paper or via audiotape. After answering these screening questions, all women will be asked standardized questions about the acceptability, safety and ease of use of the method to which they are randomized.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 or an emancipated minor

Exclusion Criteria:

* Child undergoing acute resuscitation
* Other adults in the room

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-01; Study Completion 2005-03

PRIMARY OUTCOMES:
Acceptability, perceived safety and ease of administration of each survey method

SECONDARY OUTCOMES:
Disclosure of domestic violence

CONTACTS AND LOCATIONS:
Overall Officials: Megan H Bair-Merritt, Principal Investigator — Children's Hospital of Philadelphia; Joel A Fein, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia Emergency Department, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Bair-Merritt MH, Feudtner C, Mollen CJ, Winters S, Blackstone M, Fein JA. Screening for intimate partner violence using an audiotape questionnaire: a randomized clinical trial in a pediatric emergency department. Arch Pediatr Adolesc Med. 2006 Mar;160(3):311-6. doi: 10.1001/archpedi.160.3.311. PMID 16520452